CLINICAL TRIAL: NCT03179774
Title: Endovascular Revascularization for Chronic Carotid Artery Occlusion Trial (ERCAO Trial) Part 1: Prospective Clinical Registry Study Part 2: Prospective Randomized Control Trial Study
Brief Title: Endovascular Revascularization for Chronic Carotid Artery Occlusion Trial
Acronym: ERCAO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201702049RINA
Record Dates: First submitted 2017-05-28; First posted 2017-06-07 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Carotid Occlusion

STUDY DESIGN:
Intervention Model Description: Part 1: Clinical registry study (Optimal medical therapy group vs. Endovascular revascularization and optimal medical therapy) Part 2: Randomized control trial (Optimal medical therapy group vs. Endovascular revascularization and optimal medical therapy)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Clinical registry-ER and OMT (Experimental): In clinical registry setting, participants who selected Endovascular revascularization and optimal medical therapy as the treatment for carotid artery occlusion are enrolled.
  Interventions: Device: Endovascular revascularization
- Clinical registry-OMT (No Intervention): In clinical registry setting, participants who selected optimal medical therapy as the treatment for carotid artery occlusion are enrolled.
- RCT-ER and OMT (Experimental): In randomized control trial setting, participants who are randomized to received endovascular revascularization and optimal medical therapy for carotid artery occlusion are enrolled.
  Interventions: Device: Endovascular revascularization
- RCT-OMT (No Intervention): In randomized control trial setting, participants who are randomized to received optimal medical therapy for carotid artery occlusion are enrolled.

INTERVENTIONS:
Device: Endovascular revascularization — All interventions will be performed via 8F femoral sheath. Target common carotid artery will be engaged with 8F JR 4 guiding catheter. Intra-luminal wiring using coronary guidewires and microcatheters or alternative subintimal tracking with antegrade re-entry technique. Wiring would be abandoned after 30 minutes of futile effort, consumption of more than 300 ml of contrast, or when the wire tip is confirmed to be extravascular. Once wire enters distal true lumen, the microcatheter was exchanged to a 1.5 mm diameter coronary balloon for pre-dilatation. Distal embolic protection device would be deployed if an adequate landing zone can be identified. Properly sized balloon expandable stents and self-expanding stents were then deployed to scaffold the occlusion. Balloon post-dilatation may be done if stent expansion was inadequate.
  Other Names: Carotid artery stenting
  Arms: Clinical registry-ER and OMT; RCT-ER and OMT

SUMMARY:
Revascularization for carotid artery occlusion (CAO) remained controversial, there is no prospective randomized control trial (RCT) regarding carotid artery stenting (CAS) in CAO patients. The investigators conduct a prospective study composed of clinical registry arm and RCT arm. The main purpose of the study is investigate neurocognitive function at 3 months and thereafter up to 12 months.

DETAILED DESCRIPTION:
Carotid artery stenosis is an important cause of stroke. Carotid artery stenting (CAS) provides non-inferior clinical outcome comparing to carotid endarterectomy (CEA). However, revascularization for carotid artery occlusion (CAO) remained controversial, owing to failed extracranial-to-intracranial (EC-IC) artery bypass trials, anatomical hindrance for CEA, and technical limitation for CAS. In the past 10 years, the investigators devoted in endovascular therapy for CAO and published innovative and pilot study results regarding feasibility of CAS for CAO, neurocognitive function (NCF) improvement after successful CAS for CAO, and predictors for CAS success in CAO, all in high-ranking journals. Moreover, successful CAS for CAO would lead to lower mortality and stroke rate during long-term follow-up, according to the preliminary analysis from the investigators. However, there is no prospective randomized control trial (RCT) regarding CAS in CAO patients, and in fact, most of the CAS trials excluded CAO.

The investigators, with the largest volume and experience in CAO recanalization in the world, felt obliged and responsible to propose the following RCT to evaluate endovascular revascularization for chronic CAO.

The study composed of two parts. The first part composed of prospective clinical registry for CAO. The second part compose of a prospective superiority trial, rater blinded, with 1:1 randomization to evaluate the clinical efficacy of interventional therapy for CAO. Eligible candidates for CAO revealed by CT, ultrasonography, angiography, or magnetic resonance imaging (MRI), with abnormal brain perfusion demonstrated by CT perfusion study (CTP) or MRI, will be enrolled in to study. If the participants agreed for randomization, participants will be randomized into 2 groups: the optimal medical therapy (OMT) group and the endovascular revascularization plus optimal medical therapy (ER+OMT) group. The primary end-point of the trial is the NCF improvement at 3 months and thereafter up to 12 months. The secondary endpoint includes: cumulative incidence of death and stroke within 30 days after the procedure; death or ipsilateral stroke between 31 days and 1 year; major stroke, ischemic stroke, or hemorrhagic stroke within 30 days after the procedure; major stroke, ischemic stroke, or hemorrhagic stroke between 31 days and 1 year; cognitive function measured by CANTAB; change of cerebral perfusion measured by CTP; target vessel revascularization rate; technique success rate; procedure success rate; and major procedure complication.

ELIGIBILITY:
Part 1: Clinical registry study

Inclusion criteria for clinical registry study

* Patient age 20 years or older
* Abnormal cerebral perfusion by CTP or MRI
* No medical history of stroke or transient ischemic attack (TIA) ipsilateral to the carotid occlusion within 90 days of randomization
* Women must not be of childbearing potential or, if of childbearing potential, have a negative pregnancy test prior to randomization.

Exclusion Criteria for clinical registry study

* Patient has acute stroke within 90 days,
* Intolerance or allergic reaction to a study medication without a suitable management alternative.
* Patient is expected to have the ADP antagonist therapy interruption within 3 months after the procedure.
* GI hemorrhage within 1 month prior to enrollment that would preclude antiplatelet therapy
* Bleeding diathesis
* Intracranial hemorrhage within the past 12 months.
* Platelet count <100,000/μl or history of heparin-induced thrombocytopenia.
* Other high-risk cardiac sources of emboli, including left ventricular aneurysm, severe cardiomyopathy, aortic or mitral mechanical heart valve, severe calcific aortic stenosis (valve area < 1.0 cm2), endocarditis, moderate to severe mitral stenosis, left atrial thrombus, or any intracardiac mass, or known unrepaired patent foramen ovale (PFO) with prior paradoxical embolism.
* Any major surgery, major trauma, revascularization procedure within the past 1 month.
* Acute coronary syndrome within the past 1 month or acute coronary syndrome (ACS) that is not amenable to revascularization (patients should undergo planned coronary revascularization at least 30 days before randomization).
* Inability to understand and cooperate with study procedures or provide informed consent.
* Patients with < 5 years life expectancy
* Concomitant vascular conditions precluding endovascular revascularization procedure;
* Previous ipsilateral carotid artery stenting
* Intracranial aneurysm or arteriovenous malformation;
* Educational level lower than elementary school;
* Aphasia or right-sided hemiparesis
* Marked depression.
* Severe dementia.

Part 2: Randomized control study

Inclusion Criteria for randomized control study

* Patient age 20 years or older
* Abnormal cerebral perfusion by CTP or MRI
* No medical history of stroke or TIA ipsilateral to the carotid occlusion within 90 days of randomization
* Patients must have a modified Rankin Scale (mRS) ≤2 at the time of informed consent.
* Women must not be of childbearing potential or, if of childbearing potential, have a negative pregnancy test prior to randomization.
* Randomization will apply to only 1 carotid artery occlusion for patients with bilateral carotid occlusion. Intervention of the contralateral stenosis, should it exists, may be done in according to clinical indications at least 30 days prior to randomization.

Exclusion Criteria randomized control study

* Patient has acute stroke within 90 days,
* Prior major ipsilateral stroke in the past with moderate disability (mRS ≥ 3) that is likely to confound study outcomes.
* Current neurologic illness characterized by fleeting or fixed neurologic deficits that cannot be distinguished from TIA or stroke.
* Patient has significant renal insufficiency with estimated glomerular filtration rate (eGFR) <30 ml/min (at screening). and would not receive renal replacement therapy if contrast agent related nephropathy occurs
* Intolerance or allergic reaction to a study medication without a suitable management alternative.
* Patient is expected to have the ADP antagonist therapy interruption within 3 months after the procedure.
* GI hemorrhage within 1 month prior to enrollment that would preclude antiplatelet therapy
* Bleeding diathesis
* Intracranial hemorrhage within the past 12 months.
* Platelet count <100,000/μl or history of heparin-induced thrombocytopenia.
* Other high-risk cardiac sources of emboli, including left ventricular aneurysm, severe cardiomyopathy, aortic or mitral mechanical heart valve, severe calcific aortic stenosis (valve area < 1.0 cm2), endocarditis, moderate to severe mitral stenosis, left atrial thrombus, or any intracardiac mass, or known unrepaired PFO with prior paradoxical embolism.
* Major (non-carotid) surgery/procedures planned within 3 months after enrollment.
* Any major surgery, major trauma, revascularization procedure within the past 1 month.
* Acute coronary syndrome within the past 1 month or ACS that is not amenable to revascularization (patients should undergo planned coronary revascularization at least 30 days before randomization).
* Coronary artery disease with two or more proximal or major diseased coronary arteries with ≥ 70% stenosis that have not, or cannot, be revascularized.
* Inability to understand and cooperate with study procedures or provide informed consent.
* Patients with < 5 years life expectancy
* Concomitant vascular conditions precluding endovascular revascularization procedure;
* Previous ipsilateral carotid artery stenting
* Intracranial aneurysm or arteriovenous malformation;
* Educational level lower than elementary school;
* Aphasia or right-sided hemiparesis
* Marked depression.
* Severe dementia.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-05-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
NCF improvement by Alzheimer Disease Assessment Scale-Cognitive subscale (ADAS-Cog) | at 3 months and thereafter up to 12 months
  Neurocognitive function was evaluated by ADAS-Cog
NCF improvement by Mini-Mental State Examination (MMSE) | at 3 months and thereafter up to 12 months
  Neurocognitive function was evaluated by MMSE.
NCF improvement by verbal fluency test | at 3 months and thereafter up to 12 months
  Neurocognitive function was evaluated verbal fluency test
NCF improvement by verbal fluency test Color Trails Test Parts 1 | at 3 months and thereafter up to 12 months
  Neurocognitive function was evaluated by Color Trails Test Parts 1
NCF improvement by verbal fluency test Color Trails Test Parts 2 | at 3 months and thereafter up to 12 months
  Neurocognitive function was evaluated by Color Trails Test Parts 2

SECONDARY OUTCOMES:
Death and stroke | within 30 days after the procedure and between 31 days and 1 year
  Cumulative incidence of death and ipsilateral stroke
Major stroke, ischemic stroke, or hemorrhagic stroke | within 30 days after the procedure and between 31 days and 1 year
  Cumulative incidence of major stroke, ischemic stroke, or hemorrhagic stroke
Cambridge Neuropsychological Test Automated Battery (CANTAB) | at 3 months and thereafter up to 12 months
  The CANTAB is a computerized test battery for cognitive function evaluation which has been validated and widely used worldwide. CANTAB tests are simple to administer and show strong correlations to brain constructs and known deficits in various disorders, as well as high sensitivity to interventions and small changes over time. It is designed to be administered by trained psychologists with standardized procedures. Tasks of the CANTAB involving practice and attention, memory, executive function and decision making would be administered to all the participants in this study.
Change of cerebral perfusion | at 3 months and thereafter up to 12 months
  Change of cerebral perfusion measured by CT perfusion
Target vessel revascularization rate | one year
  Target vessel revascularization rate
Technique success rate | 30 days
  Technique success is defined if the occlusion segment was recanalized with final residual diameter stenosis of <20%, and establishing grade 3 antegrade Thrombolysis in Cerebral Infarction (TICI) flow.
Procedure success rate | 30 days
  Procedure success: the occlusion segment was stented with final residual diameter stenosis of <20%, and establishing grade 3 antegrade TICI flow and without periprocedural complications.

OTHER OUTCOMES:
Major procedure complication | 30 days
  Major procedure complication includes intracranial hemorrhage, myocardial infarction, embolic stroke, vascular complication and death during endovascular revascularization or within 30 days after endovascular revascularization.
Bleeding complication | one year
  any bleeding events during the study

CONTACTS AND LOCATIONS:
Overall Officials: Hsien-Li Kao, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No